CLINICAL TRIAL: NCT07017621
Title: Qualitative Study on the Experiences of Mothers 6 to 12 Months After Their Participation in the Mother-baby Groups of the HUGS Study
Acronym: HUGSquali
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/21/0166-ancillaire; 2024-A02604-43 (Other: ANSM)
Record Dates: First submitted 2025-05-20; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Postnatal Depression; Postpartum Depression (PPD)
Keywords: Postpartum Depression; mother-child interaction; early intervention; mother-baby interaction
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Mother-baby group who received the HUGS therapy

SUMMARY:
The HUGS-QUALI study is a qualitative investigation that explores the experiences of mothers who participated in HUGS mother-baby therapy groups. Conducted 6 to 12 months after the intervention, the study aims to understand how this culturally adapted therapy influences the bond between mothers and their infants and affects their daily lives. By collecting detailed personal stories through in-depth interviews, the study seeks to understand if the adapted HUGS program effectively support French mothers in improving their interactions with their babies, when facing postpartum depression.

DETAILED DESCRIPTION:
Postpartum depression affects 15-20% of women in France and is often associated with impaired mother-infant interactions, a disruption observed in up to 73% of cases that can adversely influence both short and long-term child development. Although standard treatments effectively reduce depressive symptoms, they frequently fail to enhance the quality of the maternal bond, underscoring the need for interventions specifically targeted at early relational dynamics. The HUGS program (Happiness, Understanding, Giving, and Sharing), a brief cognitive behavioral therapy originally validated by Professor Jeannette Milgrom's Australian team, has been culturally adapted for the French context to improve mother-infant relationships. The ancillary HUGS-QUALI study employs a qualitative approach by conducting in-depth interviews with mothers 6 to 12 months following their participation in HUGS mother-baby groups, implemented across several French maternity centers.

ELIGIBILITY:
Inclusion Criteria:

* Women who participated in the HUGS mother-baby groups of the HUGS study (at various recruitment sites: Toulouse University Hospital (Paule de Viguier Maternity), Joseph Ducuing Maternity in Toulouse, and Bordeaux Maternity) and who have completed their follow-up as part of the original study.

Exclusion Criteria:

* Women refusing to participate in the study.
* Women who did not participate in the HUGS group of the HUGS study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study participants are drawn from a clinical cohort of mothers who attended HUGS mother-baby groups at specialized maternity centers in France. Specifically, they represent patients from Toulouse University Hospital (Paule de Viguier Maternity), Joseph Ducuing Maternity in Toulouse, and Bordeaux Maternity. These women, must have completed the follow-up of the original HUGS study.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2026-02-04 (Estimated); Study Completion 2026-02-04 (Estimated)

PRIMARY OUTCOMES:
Qualitative Analysis of Maternal Narratives Reflecting the Impact of the Intervention on the Mother-Infant Relationship | 6 to 12 months after completion of the HUGS mother-baby therapy groups.
  Qualitative thematic analysis of interview transcripts (no specific scale nor questionnaire) the semi directive interview guideline is confidential.
  Each interview will undergo multiple readings to identify emerging themes and sub-themes. The thematic framework will be validated through coding triangulation to ensure consistency and reliability of the findings.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Paule De Viguier Hospital, Toulouse, Occitanie
  - Bordeaux Public Hospital, Bordeaux
  - Joseph Ducuing, Toulouse